CLINICAL TRIAL: NCT00710008
Title: Effect of Short-Term Exercise Training on ATP Synthesis in Relatives of Type 2 Diabetic Humans
Acronym: RECO1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Landsteiner Institut (Other)
Collaborators: Mein Hanusch-Krankenhaus (Other); Karl-Landsteiner Institute for Endocrinology and Metabolism (Unknown); Medical University of Vienna (Other); Lund University Hospital (Other); Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy (Other Government)
Responsible Party: Landsteiner Institute, Landsteiner Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCT00481598
Record Dates: First submitted 2008-06-30; First posted 2008-07-03 (Estimated); Last update posted 2008-08-20 (Estimated); Status verified 2008-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: type 2 diabetes,; exercise training,; ATP-synthesis,; intramyocellular lipids,; hepatocellular lipids; first degree relatives of; patients
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: exercise training — 3 bouts of exercise at 90%RCP during one week

SUMMARY:
First degree relatives of type 2 diabetic patients (T2DM) suffer an increased risk of developing this disease themselves, starting with impaired insulin sensitivity. This risk can be minimized by lifestyle interventions such as regular exercise training. Until this day, little is known about the short-term effects of exercise training on insulin sensitivity and the lipid content of the liver and skeletal muscle.

DETAILED DESCRIPTION:
Life style intervention including diet and exercise is the recommended strategy for the prevention of type 2 diabetes mellitus (T2DM). First-degree relatives of patients with type 2 diabetes mellitus (T2DM) have an increased risk of insulin resistance and T2DM. According to the current paradigm, inherited and environmental factors cause insulin resistance by increasing intramyocellular lipid metabolites and stimulation of inflammatory pathways which both interfere with insulin signal transduction leading to an impaired rise of glucose-6-phosphate (G6P) upon insulin stimulation indicating impaired glucose transport/phosphorylation. In sedentary humans, these alterations can coexist with excessive storage of triglycerides as intramyocellular or hepatocellular lipids (IMCL, HCL). This indicates reduction of the muscles´ oxidative capacity which has been confirmed by demonstration of decreased mitochondrial function and/or number in insulin resistant states such as aging, increased availability of plasma free fatty acids (FFA) and overt T2DM. Likewise, severely insulin resistant, but nondiabetic relatives present with elevated FFA, IMCL and HCL along with impaired mitochondrial ATP synthesis which most likely results from reduced mitochondrial contents. However, it is unclear whether these alterations are only due to inherited abnormalities of mitochondrial biogenesis or secondary to chronically impaired glucose tolerance, increased lipid availability or inflammatory processes which are controlled by cytokines such as adiponectin, visfatin and retinol binding protein-4 (RBP4).

Likewise it remains uncertain to which extent such abnormalities are reversible by physical exercise stimulation and/or occur independently of effects on insulin action.

Long-term endurance exercise training increases insulin sensitivity in sedentary young and elderly healthy, first degree relatives of type 2 diabetic patients, glucose intolerant and obese nondiabetic or type 2 diabetic humans. Exercise training for at least 4 weeks also enhances fat oxidation along with increased size, number and enzyme activities of mitochondria. However, little is known on the time course and onset of exercise-induced changes in glucose and energy metabolism independently of the acute exercise effects occurring within the first 24 hours. At 48 hours after one bout of aerobic exercise, insulin-stimulated glucose disposal and IMCL can be increased or unchanged. Effects of short-term exercise on the underlying energy generating pathways have not yet been reported in vivo in humans. Flux of inorganic phosphate (Pi) to ATP through ATP synthase (fATPase) provides a measure of mitochondrial ATP synthesis.

We use multinuclear magnetic resonance spectroscopy (MRS) to simultaneously measure fATP as well as G6P, IMCL and HCL before and after three bouts of cycling training. We will test the hypotheses that short-term exercise training simultaneously increases fATPase and insulin sensitivity in healthy humans (control) and in relatives. Furthermore, we will investigate whether baseline fATPase reflects whole-body oxidative capacity and whether post-exercise fATPase is influenced by lipid availability due to alterations in IMCL, HCL or circulating triglycerides or FFA.

ELIGIBILITY:
Inclusion Criteria:

* First degree relatives of type 2 diabetic patients
* Age: 18-50 years
* BMI <30 kg/m2 (due to limited MR diameter)
* Normal routine lab tests (blood cell count, kidney, liver, pancreas, thyroid and neuromuscular function)
* Availability within the local area throughout the study
* Ability to understand and sign the consent forms

Exclusion Criteria:

* Current smoking
* Present drug treatment
* Regular exercise training
* Contraindications for MRS studies: claustrophobia and metalliferous implants
* Pregnancy
* HIV or Hepatitis
* Acute disease 2 weeks previous to the examination
* Heart disease
* Hypertension (RR>140/95)
* Liver disease
* Kidney disease
* Pulmonary disease
* Thyroid disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-02; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
ATP-Synthesis, liver lipid content, skeletal muscle lipid content

CONTACTS AND LOCATIONS:
Overall Officials: Michael Roden, Prof.Dr., Study Director — Landsteiner Institute
Locations (1):
- Landsteiner Institute, Vienna, Vienna, Austria